CLINICAL TRIAL: NCT06311734
Title: A Single-center, Randomized, Double-blind,Placebo-controlled Study, to Evaluate Safety,Tolerability, Pharmacokinetics and Pharmacodynamics of LW231 in Healthy Volunteers and Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Study of LW231 to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Healthy Volunteers and Participants With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Longwood Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LW231-I-01
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: SAD in healthy participants (Experimental): Part A: Single ascending doses of up to 800 mg LW231 tablets in healthy participants.
  Interventions: Drug: LW231 tablets; Drug: Placebo
- Part b: MAD in healthy participants (Experimental): Part B: Multiple ascending doses of up to 400 mg LW231 tablets in healthy participants. Dosages will be determined from data collected from Part A.
  Interventions: Drug: LW231 tablets; Drug: Placebo
- Part c: MAD in CHB participants (optional) (Experimental): Part C: Multiple ascending doses of up to 400 mg LW231 tablets in CHB participants. Dosages will be determined from data collected from Part A and Part B.
  Interventions: Drug: LW231 tablets; Drug: Placebo

INTERVENTIONS:
Drug: LW231 tablets — P.O.
  Other Names: LW231
Drug: Placebo — P.O.

SUMMARY:
To Evaluate the Tolerability and Pharmacokinetics of LW231 Tablets in Single-center, Randomized, Double-blind, Placebo-controlled Multiple-dose, Single-dose, Multiple-dose Phase Ia Clinical Trials in Healthy Subjects .

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of LW231 tablets in healthy volunteers and in chronic hepatitis B (CHB) patients after single and multiple doses. In addition, the study will evaluate the initial antiviral efficacy of LW231 in CHB patients following a multiple dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

1.18-55 years old male or female. 2.Body Mass Index (BMI) between 18 to 28 kg/m2 (inclusive) and body weight equal to or over 45 kg for females and 50kg for males.

3.Healthy status will be defined as the absence of evidence of any active or chronic disease following a detailed medical and surgical history, concomitant drug use (including hormonal supplements), a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology, and urinalysis.

Exclusion Criteria:

1. Any clinically significant abnormalities in laboratory test results at screening. In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility.
2. Participants who have donated over 450 mL of blood or blood products or had significant blood loss within three months prior to screening.
3. Heavy smokers (those who smoke greater than or equal to 5 or more cigarettes a day within three months prior to screening).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 4 days for SAD, up to 3 days after the last dose of study drug for MAD
  An adverse event (AE) was defined as any untoward medical occurrence in a participant who was administered a pharmaceutical product (including investigational drug) during the course of a clinical investigation. An AE could therefore be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease that was temporally associated with the use of the investigational product, regardless of whether it was considered to be related to the investigational product or not.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of LW231 | Up to 4 days after the last dose of study drug
Time to Cmax (Tmax) of LW231 | Up to 4 days after the last dose of study drug
Area Under the Curve From Time 0 to the Last Measurable Concentration (AUClast) of LW231 | Up to 4 days after the last dose of study drug
Area Under the Curve From Time 0 to 24 Hours (AUC0-24) of LW231 | Up to 4 days after the last dose of study drug
Half-life (t1/2) of LW231 | Up to 4 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No